CLINICAL TRIAL: NCT05195164
Title: The Effects of Orchiectomy and Age on Vascular and Metabolic Health in Older Versus Younger Transgender Women
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20-2141; NIH 5 K12 HD057022 (Other Grant/Funding Number: Building Interdisciplinary Research Careers in Women's Health (BIRCWH) - K12)
Record Dates: First submitted 2021-10-22; First posted 2022-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Transgender; Gender Identity; Vascular Stiffness; Vascular Inflammation; Insulin Sensitivity; Blood Pressure; Lipid Disorder; Appetitive Behavior
MeSH Terms: conditions — Insulin Resistance; Lipid Metabolism Disorders; Appetitive Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and endothelial cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older transgender women: This cohort will consist of healthy transgender women aged 45 and above who have not undergone but desire orchiectomy, who have been on estrogen (history of oral, transdermal or injectable) and spironolactone for at least one year.
  Interventions: Other: No intervention
- Younger transgender women: This cohort will consist of healthy transgender women aged 18-44 who have not undergone but desire orchiectomy, who have been on estrogen (history of oral, transdermal or injectable) and spironolactone for at least one year.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There was no intervention

SUMMARY:
This study plans to learn more about differences in heart disease risk after gender-affirming orchiectomy (i.e., testes removal) in older transgender (trans) women compared to younger trans women.

DETAILED DESCRIPTION:
The global aim of this study is to characterize cardiometabolic risk (measured by vascular, metabolic and biochemical factors-which have not been extensively studied prospectively) in trans women before and after orchiectomy. Trans women appear to be at greater risk for cardiovascular disease (CVD) and blood clots compared to non-trans adults. The effect of orchiectomy on CVD risk among trans women is unknown, but orchiectomy may change blood vessel function and metabolic health. The investigators will examine blood vessel function and metabolic profiles of trans women before and at several timepoints after orchiectomy to identify age-related differences in CVD risk factors. This knowledge may lead to new approaches to prevent CVD in trans women as well as all people regardless of gender identity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Identify as a transgender woman
* Have taken estradiol and spironolactone for at least one year
* Currently taking oral or transdermal or injectable estradiol
* Have not yet undergone but desire orchiectomy

Exclusion Criteria:

* Under 18 years of age
* Don't identify as a transgender woman
* Not currently taking estradiol or spironolactone
* Have been on estradiol and spironolactone for less than one year
* History of orchiectomy
* Not deemed a candidate for orchiectomy
* Current tobacco smoker
* Current illicit drug use
* History of prior or active estrogen-dependent neoplasms
* Acute liver or gallbladder disease
* Venous thromboembolism
* Hypertriglyceridemia >500 mg/dL
* Fasted plasma glucose >7.0 mmol/L or previously treated diabetes
* Resting blood pressure >140/90 mmHg

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender women (people who were assigned male at birth but whose gender identity is female). They may or may not have legally changed their gender marker.
Study Population: Transgender women from the Denver metropolitan area and/or who utilize health care at University of Colorado Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of endothelial function (flow-mediated dilation (FMD) at Baseline | Baseline
  Brachial artery flow-mediated dilation (FMD), as measured by ultrasound.
Evaluation of endothelial function (flow-mediated dilation (FMD) at 1 Month | 1 month
  Brachial artery flow-mediated dilation (FMD), as measured by ultrasound.
Evaluation of endothelial function (flow-mediated dilation (FMD) at 6 Months | 6 month
  Brachial artery flow-mediated dilation (FMD), as measured by ultrasound.
Evaluation of endothelial function (flow-mediated dilation (FMD) at 12 Months | 12 month
  Brachial artery flow-mediated dilation (FMD), as measured by ultrasound.

SECONDARY OUTCOMES:
Evaluation of carotid artery compliance | Baseline, 1 mo., 6 mo., 12 mo.
  The carotid artery compliance index indicates how elastic the artery is. The index describes the change in arterial blood volume in response to a change in arterial blood pressure. Lower numbers are associated with worse outcomes (less elastic arteries).
Evaluation of carotid artery beta stiffness index | Baseline, 1 mo., 6 mo., 12 mo.
  The carotid artery beta stiffness index indicates how stiff the artery is. Higher numbers are associated with worse outcomes (stiffer artery).
Carotid artery intimal-medial thickness | Baseline, 1 mo., 6 mo., 12 mo.
Evaluation of oxidant burden: oxidized LDL | Baseline, 1 mo., 6 mo., 12 mo.
  Oxidized low-density lipoprotein (LDL) measured in the blood and endothelial cells.
Evaluation of oxidant burden: nitrotyrosine | Baseline, 1 mo., 6 mo., 12 mo.
  Nitrotyrosine measured in the blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: nuclear factor kappa-light-chain-enhancer of activated B cells (NFkB) | Baseline, 1 mo., 6 mo., 12 mo.
  Protein NFkB (nuclear factor kappa-light-chain-enhancer of activated B cells) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: MCP-1 | Baseline, 1 mo., 6 mo., 12 mo.
  Monocyte Chemoattractant Protein-1 (MCP-1) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: IL-6 | Baseline, 1 mo., 6 mo., 12 mo.
  Interleukin 6 (IL-6) measured in blood and endothelial cells.
Evaluation of vascular endothelial cell inflammation: CRP | Baseline, 1 mo., 6 mo., 12 mo.
  C-reactive protein (CRP) measured in blood and endothelial cells.
Blood pressure | Baseline, 1 mo., 6 mo., 12 mo.
  Blood pressure will be measured at baseline, 1 mo., 6 mo. 12 mo.
Plasma lipid concentrations: total cholesterol | Baseline, 1 mo., 6 mo., 12 mo.
  Total cholesterol will be determined at baseline, 1 mo., 6 mo., 12 mo.
Plasma lipid concentrations: triglycerides | Baseline, 1 mo., 6 mo., 12 mo.
  Triglycerides will be determined at baseline, 1 mo., 6 mo., 12 mo.
Insulin sensitivity | Baseline, 1 mo., 6 mo., 12 mo.
Whole body composition: Percent Lean Mass | Baseline, 6 mo., 12 mo.
  Percent lean mass will be determined using dual energy x-ray absorptiometry.
Whole body composition: Percent Fat Mass | Baseline, 6 mo., 12 mo.
  Percent fat mass will be determined using dual energy x-ray absorptiometry.
Regional body composition: Percent Lean Mass | Baseline, 6 mo., 12 mo.
  Regional percent lean mass will be determined using dual energy x-ray absorptiometry.
Regional body composition: Percent Fat Mass | Baseline, 6 mo., 12 mo.
  Regional percent fat mass will be determined using dual energy x-ray absorptiometry.
Bone density | Baseline, 12 mo.
  Bone density of femur and spine will be determined using dual energy x-ray absorptiometry.
Weight changes | Baseline, 1 mo., 6 mo., 12 mo.
  Body weight will be measured at baseline, 1 mo., 6 mo., 12 mo.
Appetite ratings | Baseline, 1 mo., 6 mo., 12 mo.
Appetite-related peptides | Baseline, 1 mo., 6 mo., 12 mo.
D-Dimer | Baseline, 1 mo., 6 mo., 12 mo.
Alcohol use | Baseline, 1 mo., 6 mo., 12 mo.
Depression symptoms | Baseline, 1 mo., 6 mo., 12 mo.
Physical activity monitoring | 7 days at baseline, 1 mo., 6 mo., 12 mo.
  Physical activity will me monitored for 7 days with an ActivPAL monitor
Energy intake | 3 days at baseline, 1 mo., 6 mo., 12 mo.
  Energy intake will be estimated with a 3-day food diary
Sex hormone concentrations | Baseline, 1 mo., 6 mo., 12 mo.
  Sex hormone concentrations of estradiol, testosterone, follicle stimulating hormone (FSH), luteinizing hormone (LH) and sex hormone-binding globulin (SHBG) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Sean Iwamoto, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No